CLINICAL TRIAL: NCT03405922
Title: Perianal Nerval Block in Proctological Interventions: a Prospective Randomized Double Blinded Study
Brief Title: Perianal Nerval Block in Proctological Interventions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Perianal block in proctology
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Perianal Fistula; Fissure in Ano; Hemorrhoids
MeSH Terms: conditions — Fissure in Ano; Hemorrhoids | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo 40 mL Saline 0.9%
  Interventions: Drug: Placebo 40 mL Saline 0.9%
- Ropivacain (Active Comparator): 40 mL Ropivacain 0.5%
  Interventions: Drug: 40 mL Ropivacain 0.5%

INTERVENTIONS:
Drug: Placebo 40 mL Saline 0.9% — Injection of 40 mL 0.9% saline
  Arms: Placebo
Drug: 40 mL Ropivacain 0.5% — Ropivacaine Hcl 0.5% Injection 40 mL
  Arms: Ropivacain

SUMMARY:
The aim of this study is to evaluate whether a local perianal block performed during a proctological intervention can reduce the postoperative pain.

DETAILED DESCRIPTION:
The aim of this study is to evaluate whether a local perianal block performed during a proctological intervention can reduce the postoperative pain.

All patients will undergo surgery under general or spinal anesthesia. At the end of the surgery, the surgeon will perform a perianal block using the local anesthetic or the placebo upon randomisation. The experimental group will receive a local anesthetics and the control group a normal saline injection. All injections will be perianal, peripheral to the external anal sphincter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with surgical indication for hemorrhoids, fistula-in-ano or anal fissures.
* Age of 18 or above

Exclusion Criteria:

* age under 18.
* Patients unable to understand an informed consent.
* Emergency operations
* Pregnant women.
* Patients with acute perianal infection.
* Patients allergic to any component of the local anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | 24 hours post-surgery
  Postoperative Pain assessed by visual analogue scale (max. 10, min.0 points, range: 0-10; 0 = no pain at all, 10 = worst pain ever experienced)

SECONDARY OUTCOMES:
Quality of Life assessed by questionnaire | 2 weeks post-surgery
  Quality of Life assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Steinemann, Principal Investigator — St:Claraspital
Locations (1):
- St Claraspital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rotigliano N, Fuglistaler I, Guenin MO, Dursunoglu GB, Freiermuth D, von Flue M, Steinemann DC. Perianal block with ropivacaine as a supplement to anaesthesia in proctological surgery: double-blind randomized placebo-controlled trial (PERCEPT). Br J Surg. 2020 Jul;107(8):960-969. doi: 10.1002/bjs.11520. Epub 2020 Mar 18. PMID 32187663